CLINICAL TRIAL: NCT01505010
Title: Investigator-Steered Project on Intravascular Renal Denervation for Management of Drug-Resistant Hypertension
Brief Title: Renal Denervation for Management of Drug-Resistant Hypertension
Acronym: INSPiRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jan A. Staessen, Professor of Medicine, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSPiRED, version 4.0
Record Dates: First submitted 2012-01-03; First posted 2012-01-06 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Treatment-resistant hypertension; Renal denervation; Sympathetic nervous system
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Parallel group trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Standard antihypertensive drug treatment
  Interventions: Procedure: Renal denervation
- Intervention group (Experimental): Renal denervation plus standard antihypertensive drug treatment
  Interventions: Procedure: Renal denervation

INTERVENTIONS:
Procedure: Renal denervation — Renal denervation in the intervention group
  Other Names: Renal denervation, using an intravascular catheter system

SUMMARY:
INSPiRED is a multicenter parallel-group trial comparing usual medical treatment (control group) or usual medical treatment plus renal denervation (intervention). In both groups adherence will be monitored both before randomization and during 36 months of follow-up.

DETAILED DESCRIPTION:
Objectives:

To compare the blood pressure lowering efficacy and safety of renal denervation vs. usual medical therapy. The primary endpoints for efficacy and safety are the baseline-adjusted between-group differences in 24-h systolic blood pressure and in glomerular filtration rate as estimated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. Secondary endpoints for efficacy and safety include other indexes of blood pressure control and renal function, metabolic variables and morbidity and mortality. These endpoints will be assessed 6 months after randomization.

Trial design:

Randomized controlled trial with blinded assessment of the primary and secondary endpoints. The study consists of 6 stages. Supervised and nonsupervised follow-up refer to assessment of outcome at or outside the participating center, respectively.

* Screening involves checking eligibility and ruling out secondary hypertension.
* Run-in period of 3 months to optimize medical treatment and to assess adherence to treatment.
* Stratification and randomization Eligible patients will be stratified by center and age group (adults vs. elderly, 20-49 vs. 50-69 years) and randomized centrally in a one-to-one proportion to control or intervention.
* Renal sympathetic denervation in the intervention group, patients of the control group will be offered renal denervation after 6 months.
* Supervised follow-up at 1, 3 and 6 months after randomization.
* Long-term supervised or non-supervised follow-up of morbidity and mortality beyond 6 months and up to 3 years.

Sample size:

To detect a 10-mm Hg difference (SD 20 mm Hg) in systolic blood pressure between the randomized groups with a 2-sided P-value of 0.01 and 90% power in total 240 patients need to be randomized. Allowing 50% screening failures, 480 patients would have to be screened.

Assessment of adherence:

Adherence to treatment will be assessed by measurement of drugs or drug metabolites in biological fluids. Jung and coworkers developed a liquid chromatography-mass spectrometric method that allows detecting all antihypertensive drugs or their metabolites in a single urine sample. This obligatory approach will be implemented.

Assessment of quality of life Assessment of quality of life is compulsory at baseline and at each visit during the supervised follow-up, using the EuroQol 5D.

Assessment of sympathetic modulation:

heart rate variability (HRV) will be assessed at baseline and at the 6-month follow-up visit, based on 15 minutes ECG recordings. A software program, developed in LabVIEW by the group of Aubert et al. will be used.

Relevance:

INSPiRED differs from previous and ongoing studies in several aspects: (1) a stringent selection of patients; (2) drug optimization with assessment of adherence throughout the study; (3) out-of-the-office blood pressure for patient selection and follow-up; (4) state-of-the-art renal artery imaging by computerized tomographic angiography; (5) validation of urinary proteomic biomarkers to predict blood pressure responses and changes in renal function; (6) follow-up will be beyond 6 months up to 3 years; (7) use of heart rate variability and renal nerve stimulation to assess the completeness of renal denervation.

ELIGIBILITY:
Inclusion criteria:

* Women and men are eligible. Women of reproductive age should apply effective contraception.
* Age ranges from 20 years (inclusive) to less than 70 years.
* Patients should have essential hypertension.
* Treatment-resistant hypertension in patients taking a stable drug regimen for at least 4 weeks consisting of 3 or more antihypertensive medications from different classes, including a diuretic.
* Under maximal therapy, office blood pressure should be ≥140/90 mmHg and the 24-h ambulatory blood pressure should be 130 mm Hg systolic or 80 mm Hg diastolic or higher.
* eGFR must be ≥ 60 mL/min/1.73 m2.
* The patients should accept to have adherence checked before randomisation and during supervised follow-up, but both patients and doctors will remain blinded to the results;
* Informed written consent.

Exclusion criteria:

* Suboptimal clinical context, because of recent history or concurrent disease.
* Isolated systolic and diastolic hypertension.
* Body-mass index ≥ 40kg/m2.
* The anatomy of the renal arteries is suboptimal for renal denervation.
* Pregnancy.
* Alcohol or substance abuse or psychiatric illnesses.
* Participation in other study.
* The clinical context is suboptimal for renal denervation.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan A. Staessen, MD, PhD, Principal Investigator — University of Leuven
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Leuven

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be made available via a motivated data transfer request (for scientific purposes only) via the PI (Prof Jan A. Staessen) and pending ethics approval.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Currently available until 2025
Access Criteria: Ethics approval

REFERENCES:
- [Result] Jacobs L, Persu A, Huang QF, Lengele JP, Thijs L, Hammer F, Yang WY, Zhang ZY, Renkin J, Sinnaeve P, Wei FF, Pasquet A, Fadl Elmula FEM, Carlier M, Elvan A, Wunder C, Kjeldsen SE, Toennes SW, Janssens S, Verhamme P, Staessen JA; European Network Coordinating Research on Renal Denervation. Results of a randomized controlled pilot trial of intravascular renal denervation for management of treatment-resistant hypertension. Blood Press. 2017 Dec;26(6):321-331. doi: 10.1080/08037051.2017.1320939. Epub 2017 May 10. PMID 28489464
- [Derived] Jin Y, Jacobs L, Baelen M, Thijs L, Renkin J, Hammer F, Kefer J, Petit T, Verhamme P, Janssens S, Sinnaeve P, Lengele JP, Persu A, Staessen JA; investigator-steered project on intravascular renal denervation for management of drug-resistant hypertension (INSPiRED) investigators. Rationale and design of the Investigator-Steered Project on Intravascular Renal Denervation for Management of Drug-Resistant Hypertension (INSPiRED) trial. Blood Press. 2014 Jun;23(3):138-46. doi: 10.3109/08037051.2014.899297. Epub 2014 Apr 17. PMID 24742341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 28 March 2014 until 11 May 2016, 3 Belgian centers screened 29 patients, of whom 4 did not meet the criteria to enter the run-in period. Of 25 remaining patients, 8 were not eligible for randomization. Of 17 eligible patients, 9 were randomized to control and 8 to RDN. Of the 8 patients randomized to intervention, two did not undergo RDN.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 9 | 8
Completed | 9 | 6
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treatment resistant hypertensive patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (8.8) | 48.4 (10.8) | 48.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Baseline to 6 Months on 24-h Ambulatory Measurement (Follow-up Minus Baseline Measurement)
Description: The primary endpoint deals with efficacy of renal denervation with regard to controlling blood pressure on ambulatory measurement. It consists of the baseline-adjusted between-group difference in the changes in 24-h systolic blood pressure. Because automated blood pressure monitors will be used, the assessment of the primary endpoint is blind.
Time Frame: The primary endpoint has been assessed 6 months after randomization.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 9 | 6
mmHg | 0.7 [-12.0 to 13.4] | -21.7 [-33.4 to -9.9]
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; We used mixed models to compare blood pressure changes between randomized groups at 6 months, while adjusting for the baseline blood pressure; statistical significance was a P-value less than 0.05 on two-sided tests; Test type: Superiority; p = 0.018, Mixed Models Analysis; Adjusted for the baseline 24-h systolic blood pressure; Mean Difference (Final Values) = 22.4, Standard Error of Mean 8.5 — Difference at 6 months in 24-h systolic blood pressure (control minus intervention)

2. Primary Outcome: Change in Glomerular Filtration Rate
Description: The primary endpoint for safety of renal denervation is the baseline-adjusted between group difference in the change of glomerular filtration rate estimated by using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation.
Time Frame: This endpoint has been assessed 6 months after randomization.
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m2
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 9 | 6
ml/min/1.73 m2 | 81.6 (24.1) | 92.4 (15.9)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Difference between control and intervention group at 6 months; Test type: Superiority or Other; p = 0.86, t-test, 2 sided; Mean Difference (Net) = 2.5, Standard Error of Mean 4.87

3. Secondary Outcome: The Intensity of Medical Treatment
Description: The number and doses of blood-pressure lowering drugs in the 2 arms of the trial.
Time Frame: This endpoint will be assessed 6 months after randomization.
Measure: Median (Inter-Quartile Range); unit: number of drugs taken per day
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 9 | 6
number of drugs taken per day | 4 [4 to 6] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Wilcocon rank sum test; Test type: Superiority; p = 0.032, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.7
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.7, Standard Error of Mean 0.8

ADVERSE EVENTS:
Time Frame: 6 months
Description: Follow-up at participating clinical centers.
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6

LIMITATIONS AND CAVEATS:
Ethical approval was obtained to randomise 18 patients in a pilot trial, published recently (http://dx.doi.org/10.1080/08037051.2017.1320939)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No